CLINICAL TRIAL: NCT00393328
Title: Bioequivalence Study of Atazanavir Single 300 mg Capsule Relative to Two Atazanavir 150 mg Capsules in Healthy Subjects
Brief Title: Bioequivalence Study of Atazanavir 300 mg Capsule
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AI424-282
Record Dates: First submitted 2006-10-23; First posted 2006-10-27 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2008-06

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — atazanavir, ritonavir drug combination; Aripiprazole

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Atazanavir + Ritonavir
- B (Active Comparator)
  Interventions: Drug: Atazanavir + Ritonavir

INTERVENTIONS:
Drug: Atazanavir + Ritonavir — Capsules, Oral, ATV 300mg as 2-150mg + RTV 100mg, single dose, 7 days washout crossed over to Treatment B.
  Other Names: Abilify
  Arms: A
Drug: Atazanavir + Ritonavir — Capsules, Oral, ATV 300mg as single cap + RTV 100mg, single dose, 7 days washout.
  Other Names: Abilify
  Arms: B

SUMMARY:
The purpose of this clinical research study is to assess the bioequivalence of atazanavir administered as a single 300 mg capsule relative to two atazanavir 150 mg capsules in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between the ages of 18 to 50 years old with a body mass index (BMI) of 18 to 30 kg/m²
* Prior to enrollment, subjects must have physical and laboratory test findings within normal limits, and women of childbearing potential (WOCBP) must have a negative pregnancy test.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46
Dates: Start 2006-11; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Blood atazanavir pharmacokinetic sampling to be collected on days 1, 2 and 3 of each of the 2 periods of the study

SECONDARY OUTCOMES:
Blood ritonavir pharmacokinetic sampling to be collected on days 1, 2 and 3 of each of the 2 periods of the study
Safety parameters including physical exam (PE), vital signs (VS), electrocardiogram (ECG) and clinical laboratory tests will be collected at study discharge

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Hamilton, New Jersey, United States